CLINICAL TRIAL: NCT04578717
Title: Effect of Surface Pre-conditioning With Bioactive Glass Air-abrasion on the Clinical Performance of Composite Restorations in Non-carious Cervical Lesions
Brief Title: Bioactive Glass Air-abrasion and Non-carious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3479-2018
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cervical Lesion
Keywords: Non-carious cervical lesions (NCCLs); Air-abrasion; Bioactive glass; Composite restorations; Adhesive
MeSH Terms: interventions — Air Abrasion, Dental

STUDY DESIGN:
Intervention Model Description: A hundred teeth with NCCLs meeting the inclusion criteria were randomly assigned into four experimental groups (n=25); A: air-abrasion + Etch&rinse, B: air-abrasion + Self-etch, C: Etch&rinse and D: Self-etch.
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical evaluation of NCCLs restorations was conducted by two trained and calibrated examiners.The examiners and patients were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Air-abrasion + Etch & rinse adhesive (Experimental): Air-abrasion unit was used to pre-condition the NCCLs with bioactive glass 45S5 followed by etch&rinse adhesive application using 37% Phosphoric acid for 30 sec and 15 sec respectively. NCCLs were rinsed thoroughly for 20 sec to remove the acid. Excess water was removed using a cotton pellet to leave a moist dentine surface. One coat of bonding adhesive was gently scrubbed on the entire enamel and dentin surface for 20 sec, air dried for 5 sec and light cured for 10 sec using LED curing light
  Interventions: Procedure: Air-abrasion; Procedure: Adhesive application - Etch&rinse
- Air-abrasion + Self-etch adhesive (Experimental): Air-abrasion unit was used to pre-condition the NCCLs with bioactive glass 45S5 followed by self-etch adhesive application which was applied to enamel and dentine for 20 sec with agitation, gently air dried and light cured for 10 sec.
  Interventions: Procedure: Air-abrasion; Biological: Adhesive application - Self-etch
- Etch & rinse adhesive (Experimental): Enamel and dentine were etched using 37% Phosphoric acid for 30 sec and 15 sec respectively. NCCLs were rinsed thoroughly for 20 sec to remove the acid. Excess water was removed using a cotton pellet to leave a moist dentine surface. One coat of bonding adhesive was gently scrubbed on the entire enamel and dentin surface for 20 sec, air dried for 5 sec and light cured for 10 sec using LED curing light
  Interventions: Procedure: Adhesive application - Etch&rinse
- Self-etch adhesive (Experimental): The bonding adhesive was applied to enamel and dentine for 20 sec with agitation, gently air dried and light cured for 10 sec.
  Interventions: Biological: Adhesive application - Self-etch

INTERVENTIONS:
Procedure: Air-abrasion — A clinical air-abrasion unit was used to pre-condition the NCCLs with bioactive glass 45S5 powder for 10 sec. The operating parameters were; air pressure, 20 psi; powder particles size, 20 µm; nozzle angle, 90◦; nozzle-lesion distance, 5 mm and the internal nozzle diameter, 900 µm
  Other Names: surface pre-conditioning
  Arms: Air-abrasion + Etch & rinse adhesive; Air-abrasion + Self-etch adhesive
Procedure: Adhesive application - Etch&rinse — Enamel and dentine were etched using 37% Phosphoric acid for 30 sec and 15 sec respectively. NCCLs were rinsed thoroughly for 20 sec to remove the acid. Excess water was removed using a cotton pellet to leave a moist dentine surface. One coat of bonding adhesive was gently scrubbed on the entire enamel and dentin surface for 20 sec, air dried for 5 sec and light cured for 10 sec using LED curing light. The light intensity of curing unit was calibrated daily using curing radiometer .
  Other Names: Bonding
  Arms: Air-abrasion + Etch & rinse adhesive; Etch & rinse adhesive
Biological: Adhesive application - Self-etch — The bonding adhesive was applied to enamel and dentine for 20 sec with agitation, gently air dried and light cured for 10 sec.
  Other Names: Bonding
  Arms: Air-abrasion + Self-etch adhesive; Self-etch adhesive

SUMMARY:
Evaluating the clinical behavior of composite restorations in NCCLs when the surface is pre-conditioned using bioactive glass air-abrasion has not been reported in the dental literature. This double-blinded randomised clinical trial evaluated the effect of surface pre-conditioning with bioactive air-abrasion on the performance of composite restorations in NCCLs placed using etch&rinse and self-etch adhesive systems.

DETAILED DESCRIPTION:
15 Patients with 100 teeth meeting the inclusion criteria were enrolled in this study. NCCLs characteristics were evaluated and recorded before the placement of restorations. The cavity dimensions in millimeters (height, width, and depth), the cavity geometry (labeled at >45°, 45° - 90°, 90° - 135°, and <135°), the degree of dentin sclerosis , the existence of attrition facets, and the existence of spontaneous sensitivity were measured and recorded in the patient's form. The preoperative sensitivity was also evaluated by applying air from a dental syringe placed 2 cm from the tooth surface for 10 seconds.

NCCLs meeting the inclusion criteria were randomly assigned into four experimental groups (n=25); A: air-abrasion + etch&rinse, B: air-abrasion + self-etch, C: etch&rinse and D: self-etch.

Prophylaxis was conducted using a rubber cup with pumice and water. The color of the composite was selected using VITA classical shade guide before applying local anesthesia with Lidocaine 2% with 1:100000 adrenaline. Retraction chord was inserted into the gingival sulcus with the aid of a blunt spatula without excessive pressure to the periodontium. Teeth were isolated with rubberdam. No preparation or beveling of cavosurface margins was performed to the NCCLs.

In air-abrasion groups, a clinical air-abrasion unit was used to pre-condition the NCCLs with bioactive glass 45S5 powder for 10 sec. The operating parameters were; air pressure, 20 psi; powder particles size, 20 µm; nozzle angle, 90◦; nozzle-lesion distance, 5 mm and the internal nozzle diameter, 900 µm

For the etch&rinse groups, enamel and dentine were etched using 37% Phosphoric acid for 30 sec and 15 sec respectively. NCCLs were rinsed thoroughly for 20 sec to remove the acid. Excess water was removed using a cotton pellet to leave a moist dentine surface. One coat of bonding adhesive was gently scrubbed on the entire enamel and dentin surface for 20 sec, air dried for 5 sec and light cured for 10 sec using LED curing light ( output >800mW/cm2).

In self-etch groups, the bonding adhesive was applied to enamel and dentine for 20 sec with agitation, gently air dried and light cured for 10 sec.

NCCLs were restored using FiltekTM Z250 XT resin composite, placed in 2 mm increments and light cured for 20 s per increment. Final contour was achieved with a fine diamond rotary instrument followed by finishing and polishing using Optrapol polishing kit .

Clinical evaluation was conducted by two trained and calibrated examiners. The examiners and patients were blinded to the group assignment, in accordance with the double-blinding randomized clinical trial design. Each restoration was evaluated at baseline (one week after restoration placement), 3 months and 6 months. This evaluation was conducted according to World Federation criteria (FDI)

ELIGIBILITY:
Inclusion Criteria:

* Be at least 19 years old, be in good general and oral health and be available for follow-up visits
* NCCLs inclusion criteria are; at least 1 mm deep, involving enamel and dentin of vital teeth.

Exclusion Criteria:

* Chronic therapeutic drug history, rampant uncontrolled caries, periodontal disease, pregnancy or lactation, orthodontic appliance use, evidence of xerostomia, evidence of severe bruxing, clenching or TMD, and known sensitivity to acrylates or related materials.
* NCCLs exclusion criteria are; teeth with periapical pathology, symptoms of pulpal pathology, non-vital or previous root canal therapy, previous pulp capping and tooth hypersensitivity

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Restoration Retention Rate and Integrity | Baseline (one week after restoration placement), Change from Baseline rate of retention at 3 months, Change from Baseline rate of retention at 6 months
  The unabbreviated scale title: Restoration Retention Rate and Integrity Scale
  The minimum and maximum values: 1, 5
  Higher scores mean a worse outcome.
  1. Restoration retained, no fractures/ cracks
  2. Small hairline crack
  3. Two or larger hairline cracks and/or chipping (not affecting the marginal integrity)
  4. Chipping fractures which damage marginal quality
  5. Partial or complete loss of restoration

SECONDARY OUTCOMES:
Change in Marginal Adaptation | Baseline (one week after restoration placement), Change from Baseline marginal adaptation at 3 months, Change from Baseline marginal adaptation at 6 months
  1. Harmonious outline, no gaps, no discoloration 2.1 Marginal gap (50 µm). 2.2 Small marginal fracture. 3.1 Gap <150 µm not removable 3.2 Several small enamel or dentin fractures 4.1 Gap >250 µm or dentin/base exposed. 4.2 chip fracture damaging margins 4.3 Notable enamel or dentin wall fracture 5. Filing is loose but in situ
Change in Postoperative Hypersensitivity | Baseline (one week after restoration placement), Change from Baseline postoperative hypersensitivity at 3 months, Change from Baseline postoperative hypersensitivity at 6 months
  This will be assessed using Dentine Hypersensitivity Scale difference from the baseline values. Tooth sensitivity score was assessed by applying air from a dental syringe placed 2-cm from the tooth surface for 10 seconds.
  The unabbreviated scale title: Dentine Postoperative Hypersensitivity Scale
  The minimum and maximum values: 1, 5
  Higher scores mean a worse outcome.
  1. Subject does not respond to air stimulus,
  2. Low hypersensitivity for a limited period of time,
  3.1. Premature / slightly more intense
  3.2. Delayed/weak sensitivity; no subjective complaints, no treatment needed.
  4.1. Premature/ very intense
  4.2. Extremely delayed/weak with subjective complaints
  4.3. Negative Sensitivity Intervention necessary but not replacement.
  5. Very intense, acute pulpitis or non-vital. Endodontic treatment is necessary and restoration has to be replaced.
Change in Recurrence of Caries | Baseline (one week after restoration placement), Change from Baseline recurrence of caries at 3 months, Change from Baseline recurrence of caries at 6 months
  1. No secondary or primary caries 2. Very small and localized demineralization. No operative treatment required 3. Larger areas of demineralization, but only preventive measures necessary (dentin not exposed) 4. Caries with cavitation (localized and accessible and can be repaired) 5. Deep secondary caries or exposed dentin that is not accessible for repair of restoration
Change in Marginal Staining | Baseline (one week after restoration placement), Change from Baseline staining margin at 3 months, Change from Baseline staining margin at 6 months
  The unabbreviated scale title: Marginal Staining Scale
  The minimum and maximum values: 1, 5
  Higher scores mean a worse outcome.
  1. No marginal staining
  2. Minor marginal staining, easily removable by polishing
  3. Moderate marginal staining, not esthetically unacceptable
  4. Pronounced marginal staining; major intervention necessary for improvement
  5. Deep marginal staining not acceptable for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hussam Milly, Phd, Study Director — Damascus University
Locations (1):
- Restorative Dentistry, Faculty of Dental Medicine, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanatta RF, Silva TM, Esper M, Bresciani E, Goncalves S, Caneppele T. Bonding Performance of Simplified Adhesive Systems in Noncarious Cervical Lesions at 2-year Follow-up: A Double-blind Randomized Clinical Trial. Oper Dent. 2019 Sep/Oct;44(5):476-487. doi: 10.2341/18-049-C. Epub 2019 Jan 31. PMID 30702405
- [Background] Lawson NC, Robles A, Fu CC, Lin CP, Sawlani K, Burgess JO. Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. J Dent. 2015 Oct;43(10):1229-34. doi: 10.1016/j.jdent.2015.07.009. Epub 2015 Jul 29. PMID 26231300
- [Background] Hafer M, Jentsch H, Haak R, Schneider H. A three-year clinical evaluation of a one-step self-etch and a two-step etch-and-rinse adhesive in non-carious cervical lesions. J Dent. 2015 Mar;43(3):350-61. doi: 10.1016/j.jdent.2014.12.009. Epub 2014 Dec 23. PMID 25541248
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645
- [Background] Paula EA, Tay LY, Kose C, Mena-Serrano A, Reis A, Perdigao J, Loguercio AD. Randomized clinical trial of four adhesion strategies in cervical lesions: 12-month results. Int J Esthet Dent. 2015 Spring;10(1):122-145. PMID 25625130
- [Background] Schroeder M, Correa IC, Bauer J, Loguercio AD, Reis A. Influence of adhesive strategy on clinical parameters in cervical restorations: A systematic review and meta-analysis. J Dent. 2017 Jul;62:36-53. doi: 10.1016/j.jdent.2017.05.006. Epub 2017 May 8. PMID 28495559
- [Background] van Dijken JW. Clinical evaluation of three adhesive systems in class V non-carious lesions. Dent Mater. 2000 Jul;16(4):285-91. doi: 10.1016/s0109-5641(00)00019-1. PMID 10831784
- [Background] Loguercio AD, Luque-Martinez IV, Fuentes S, Reis A, Munoz MA. Effect of dentin roughness on the adhesive performance in non-carious cervical lesions: A double-blind randomized clinical trial. J Dent. 2018 Feb;69:60-69. doi: 10.1016/j.jdent.2017.09.011. Epub 2017 Sep 27. PMID 28962842
- [Background] Sauro S, Watson TF, Thompson I, Banerjee A. One-bottle self-etching adhesives applied to dentine air-abraded using bioactive glasses containing polyacrylic acid: an in vitro microtensile bond strength and confocal microscopy study. J Dent. 2012 Nov;40(11):896-905. doi: 10.1016/j.jdent.2012.07.004. Epub 2012 Jul 20. PMID 22819812